CLINICAL TRIAL: NCT02922023
Title: Management of Uncontrolled Hypertension: Ambulatory Blood Pressure Monitoring and Subsequent Modification of Therapy or Shifting Anti-hypertensive Medication to Night-time Dosing
Brief Title: Management of Uncontrolled Hypertension (HTN)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subjects lost to follow-up
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601421
Record Dates: First submitted 2016-09-30; First posted 2016-10-03 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Chronotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Chronotherapy (Active Comparator): Chronotherapy group automatically receives a shift in 1 anti-hypertensive medication to night-time without assessment of ambulatory blood pressure monitor results.
  Interventions: Other: Chronotherapy
- ABPM (Active Comparator): ABPM group will have their ambulatory blood pressure monitor results reviewed prior to deciding to change regimen.
  Interventions: Device: Ambulatory blood pressure monitor (ABPM)

INTERVENTIONS:
Device: Ambulatory blood pressure monitor (ABPM) — ABPM allows providers to obtain blood pressure readings over a 24 hour period, to assess blood pressure at night to determine "dipping" status, and to evaluate the efficacy of anti-hypertensive therapy.
  Arms: ABPM
Other: Chronotherapy — Chronotherapy group will receive a shift in the timing of one of their antihypertensive medications to nighttime dosing without consulting their ABPM results.
  Arms: Chronotherapy

SUMMARY:
In this study, investigators will compare chronotherapy to ABPM. Data collected will include hypertension drug therapy regimen prior to and during the study, timing of medication administration, and dose, along with the patient's office blood pressure values prior to study and one month after modification in therapy. This will enable us to explore whether it is a practical endeavor to implement ABPM as a routine process for all uncontrolled hypertension patients or whether ABPM does not seem to provide considerable value over shifting the timing of drug administration.

DETAILED DESCRIPTION:
Investigators propose to conduct a pilot study to determine whether the incorporation of Ambulatory Blood Pressure Monitoring (ABPM) as routine procedure in clinic for uncontrolled hypertension influences how anti-hypertensive drug therapy is modified or if simply shifting the dosing of anti-hypertensive medications to night time achieves similar results. Investigators will enroll 20 participants with uncontrolled hypertension, who are prescribed 3 anti-hypertensive medications at maximum dose. All twenty patients will undergo 24-hour blood pressure monitoring with ABPM at baseline and one month after change in therapy has been initiated; ten of the patients will be randomized to receive a shift in dosing schedule of anti-hypertensive medication to night-time without utilizing their ABPM results while the remaining ten will receive modifications in therapy based on their ABPM results and dipping status. The results of this study will assist in assessing the feasibility and benefits of the incorporation of ABPM into the routine management of hypertension.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years
2. Blood pressure of >130/80 mmHg
3. Currently receiving 3 anti-hypertensive agents, one of which is a diuretic, for at least six weeks

Exclusion criteria

1. Vulnerable populations

1. Pregnant women
2. Prisoners
3. Cognitively impaired persons
4. Economically and/or educationally disadvantaged
5. Human fetuses and neonates
6. Patients who work night-shift
7. Children
8. Conditions with visual field deterioration (Anterior Ischemic Optic Neuropathy, Glaucoma, Optic Nerve Disorders)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Vogel Anderson, Pharm D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronotherapy | ABPM
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: 1. Age ≥ 18 years
  2. Blood pressure of >130/80 mmHg
  3. Currently receiving 3 anti-hypertensive agents, one of which is a diuretic, for at least six weeks
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronotherapy | ABPM | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (5.5) |  | 71.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Changes in Blood Pressure
Description: changes in blood pressure from baseline vs after 1 month of change in drug therapy for each patient. Measured by T-test
Time Frame: Changes between Baseline and 1 month
Population: Data were not collected for either subject as they both withdrew from the study.
Arm/Group | Chronotherapy | ABPM
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Amount of Subjects From Each Group That Achieved Blood Pressure Goal
Description: Measured using Chi-square test or Fisher's Exact Test
Time Frame: 1 month
Population: Data were not collected for either subject as they both withdrew from the study.
Arm/Group | Chronotherapy | ABPM
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: 2 subjects were enrolled; however, they did not complete the study so no adverse events occured
Arm/Group | Chronotherapy | ABPM
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT02922023/Prot_SAP_000.pdf